CLINICAL TRIAL: NCT02051309
Title: Phase-II Clinical Trial Evaluating Guanfacine for Smoking Cessation
Brief Title: Guanfacine Clinical Trial for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1110009133_B; R01DA035001 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-01-31 (Estimated); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Smoking Cessation
Keywords: Smokers; Quit Smoking; Treatment; Guanfacine
MeSH Terms: conditions — Smoking Cessation | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Guanfacine 6mg/day ER (Experimental): Guanfacine 6mg/day extended release
  Interventions: Drug: Guanfacine
- Placebo (Placebo Comparator): Placebo matching capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine — 6mg/day ER with 3-week lead-in period. Maintained at steady state throughout 8 week treatment phase. After treatment phase, given taper supply of medication. Follow up at 1 month, 2 months and 6 months.
  Other Names: Intuniv
  Arms: Guanfacine 6mg/day ER
Drug: Placebo
  Arms: Placebo

SUMMARY:
Adult daily smokers motivated to quit smoking will be randomized to extended-release guanfacine (6mg/day) or placebo and will enroll in an 8-week treatment period combining medication with brief behavioral support. The investigators hypothesize that the active dose of guanfacine compared to placebo will increase rates of prolonged smoking abstinence at the end of the 8-week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Able to read, write and comprehend English
* Smoker
* Able to take oral medications and willing to adhere to a medication regimen
* Provide evidence of a stable living residence in the last 2 months, have reasonable transportation to the study site, and have no plans to move within the next 3 months or unresolved legal problems

Exclusion Criteria:

* Any significant current medical conditions that would contraindicate smoking
* Current Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) abuse or dependence of other substances, other than nicotine dependence or alcohol abuse
* Positive test results at intake appointment on urine drug screen for illicit drugs
* Past 30 days use of any psychoactive drugs including anxiolytics and antidepressants
* Women who are pregnant or nursing
* Suicidal, homicidal or evidence of current mental illness such as schizophrenia, bipolar disorder or major depression, or anxiety disorders
* Meeting DSM-IV criteria for current attention deficit hyperactivity disorder (ADHD)
* Individuals who are currently taking medications known to be effective for smoking cessation or are regular users of other tobacco products in the past 30 days
* Only one member per household can participate in the study
* Specific exclusions for administration of guanfacine not already specified include:
* EKG evidence at baseline screening for any clinically significant conduction abnormalities or arrhythmias
* Known intolerance for guanfacine or any alpha blocker
* History of fainting, syncopal attacks
* Heart failure or myocardial infarction
* Impaired liver (as indicated by aspartate aminotransferase (AST), alanine aminotransferase (ALT) >3x normal)
* Renal function (as indicated by estimated creatinine clearance <60cc/min)
* Treatment with any antihypertensive drug or any alpha-adrenergic blocker
* Use of any central nervous system depressant (e.g., phenothiazines, barbiturates, benzodiazepines)
* Use of strong cytochrome P450 3A4 (CYP3A4) inhibitors (e.g., ketoconazole) or inducers (e.g., rifampin), or consumption of grapefruit juice
* Subjects may not have donated blood in the past 8 weeks or have been involved in other investigational studies that involve substantial blood draws or medications unknown to us

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-03; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigations, Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Guanfacine 6mg/Day ER: Guanfacine 6mg/day extended release
  Guanfacine: 6mg/day ER with 3-week lead-in period. Maintained at steady state throughout 8 week treatment phase. After treatment phase, given taper supply of medication.
- Placebo: Placebo matching capsule
  Placebo
Period: Overall Study
Arm/Group | Guanfacine 6mg/Day ER | Placebo
Started | 58 | 63
Completed | 26 | 35
Not Completed | 32 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guanfacine 6mg/Day ER | Placebo | Total
Number analyzed (Participants) | 58 | 63 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.17 (11.70) | 47.68 (11.42) | 47.91 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 28 | 33 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 42 | 46 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 18.21 (7.67) | 18.32 (8.66) | 18.26 (8.19)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Prolonged Smoking Abstinence
Description: Prolonged smoking abstinence defined as no relapse in week 3 to week 8, in participants with available outcome data during weeks 3 to 8.
Time Frame: Week 3 to week 8 during 8-week treatment phase
Population: Participants with available outcome data during weeks 3 to 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Guanfacine 6mg/Day ER | Placebo
Number analyzed (Participants) | 31 | 40
Participants | 11 | 7

ADVERSE EVENTS:
Time Frame: During 8-week treatment period.
Arm/Group | Guanfacine 6mg/Day ER | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/63
Other Adverse Events (participants affected / at risk) | 0/58 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT02051309/Prot_SAP_000.pdf